CLINICAL TRIAL: NCT00028990
Title: A Randomized Phase III Tial Of Paclitaxel Versus Paclitaxel Plus Bevacizumab (rhuMAb VEGF) As First-Line Therapy For Locally Recurrent or Metastatic Breast Cancer
Brief Title: Paclitaxel With or Without Bevacizumab in Treating Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); NCIC Clinical Trials Group (Network); NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069156; E2100; NCCTG-E2100; CAN-NCIC-MAC3; NSABP-E2100
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel + Bevacizumab (Active Comparator)
  Interventions: Drug: bevacizumab; Drug: Paclitaxel
- Paclitaxel (Active Comparator)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: bevacizumab — 10 mg/kg following paclitaxel treatment on weeks 1 and 3 of every 4-week cycle
  Other Names: Avastin
  Arms: Paclitaxel + Bevacizumab
Drug: Paclitaxel — 90 mg/m2 IV infusion over 1 hour every week for 3 weeks followed by 1 week rest

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. It is not yet known whether paclitaxel works better with or without bevacizumab in treating breast cancer.

PURPOSE: This randomized phase III trial is to see if paclitaxel works better with or without bevacizumab in treating patients who have locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to treatment failure in patients with locally recurrent or metastatic breast cancer treated with paclitaxel with or without bevacizumab.
* Compare the objective response rate, duration of response, overall survival, and time to progression in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to disease-free interval (no more than 24 months vs more than 24 months), number of metastatic sites (less than 3 vs 3 or more), treatment with prior adjuvant chemotherapy (yes vs no), and estrogen receptor status (positive vs negative vs unknown). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 followed by bevacizumab IV over 30-90 minutes on days 1 and 15.
* Arm II: Patients receive paclitaxel as in arm I. In both arms, courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and on day 1 of weeks 17 and 33.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 316-650 patients (158-325 per treatment arm) will be accrued for this study within 31 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast
* Locally recurrent disease that is not amenable to surgical resection with curative intent OR
* Metastatic disease
* No HER-2-overexpressing (3+) breast cancer unless previously treated with trastuzumab (Herceptin)

  * Unknown HER-2 status allowed provided herceptin-based therapy inappropriate or not indicated
* No prior or radiologic evidence of CNS metastases, including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement by head CT scan or MRI
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding diathesis

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal (ULN) (5 times ULN for known liver involvement)
* PT/PTT no greater than 1.5 times normal
* INR no greater than 1.5 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* No proteinuria by dipstick urinalysis
* Trace proteinuria allowed
* Proteinuria less than 500 mg by 24-hour urine collection if proteinuria at least 1+ by urinalysis

Cardiovascular:

* No clinically significant cardiovascular disease
* No myocardial infarction within the past 12 months
* No unstable angina
* No prior deep vein thrombosis
* No grade 2 or greater peripheral vascular disease
* No uncontrolled congestive heart failure
* No uncontrolled hypertension (systolic blood pressure greater than 170 mmHg and diastolic blood pressure greater than 95 mm Hg)
* No prior cerebrovascular accident

Pulmonary:

* No prior pulmonary embolism

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* No history of seizures
* No non-healing wound or fracture
* No hypersensitivity to paclitaxel, Cremophor EL, Chinese hamster ovary cell products, or other recombinant human antibodies
* No active infection requiring parenteral antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* No prior chemotherapy for locally recurrent or metastatic breast cancer
* At least 12 months since prior adjuvant or neoadjuvant taxane therapy
* At least 3 weeks since prior adjuvant chemotherapy

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy for locally recurrent or metastatic breast cancer

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No prior radiotherapy to only site of disease
* No concurrent local radiotherapy for pain control or life-threatening situations (e.g, superior vena cava syndrome, spinal cord compression, or CNS metastases)

Surgery:

* At least 4 weeks since prior major surgical procedure except placement of vascular access device or breast biopsy
* At least 7 days since prior minor surgical procedure, including placement of an access device or fine needle aspiration

Other:

* At least 10 days since prior anticoagulant therapy (low-dose anticoagulant therapy to maintain patency of a vascular access device allowed)
* At least 10 days since prior and no concurrent daily aspirin (more than 325 mg/day) or other non-steroidal anti-inflammatory medication known to inhibit platelet function
* No concurrent dipyridamole, ticlopidine, clopidogrel, or cilostazol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2002-01-29 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | Assessed every 3 months for 2 years, then every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center; Robin Zon, MD — Elkhart General Hospital; Edith A. Perez, MD, Study Chair — Mayo Clinic; Tamara N. Shenkier, MD, Study Chair — British Columbia Cancer Agency; Melody A. Cobleigh, MD, Study Chair — Rush University Medical Center
Locations (30):
- United States (28):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Background] Gray R, Giantonio BJ, O'Dwyer PJ, et al.: The safety of adding angiogenesis inhibition into treatment for colorectal, breast, and lung cancer: the Eastern Cooperative Oncology Group's (ECOG) experience with bevacizumab (anti-VEGF). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-825, 2003.
- [Result] Schneider BP, Wang M, Radovich M, Sledge GW, Badve S, Thor A, Flockhart DA, Hancock B, Davidson N, Gralow J, Dickler M, Perez EA, Cobleigh M, Shenkier T, Edgerton S, Miller KD; ECOG 2100. Association of vascular endothelial growth factor and vascular endothelial growth factor receptor-2 genetic polymorphisms with outcome in a trial of paclitaxel compared with paclitaxel plus bevacizumab in advanced breast cancer: ECOG 2100. J Clin Oncol. 2008 Oct 1;26(28):4672-8. doi: 10.1200/JCO.2008.16.1612. PMID 18824714
- [Result] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Result] Cella D, Wang M, Wagner L, Miller K. Survival-adjusted health-related quality of life (HRQL) among patients with metastatic breast cancer receiving paclitaxel plus bevacizumab versus paclitaxel alone: results from Eastern Cooperative Oncology Group Study 2100 (E2100). Breast Cancer Res Treat. 2011 Dec;130(3):855-61. doi: 10.1007/s10549-011-1725-6. Epub 2011 Aug 27. PMID 21874312
- [Result] Miller KD, Wang M, Gralow J, et al.: A randomized phase III trial of paclitaxel versus paclitaxel plus bevacizumab as first-line therapy for locally recurrent or metastatic breast cancer: a trial coordinated by the Eastern Cooperative Oncology Group (E2100). [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-3, 2005.
- [Result] Miller KD. E2100: a phase III trial of paclitaxel versus paclitaxel/bevacizumab for metastatic breast cancer. Clin Breast Cancer. 2003 Feb;3(6):421-2. doi: 10.3816/CBC.2003.n.007. No abstract available. PMID 12636887